CLINICAL TRIAL: NCT00634907
Title: Prospective CYP2C9 And VKORC1 Genotyping For Total Hip or Knee Replacement Patients Receiving Warfarin (Coumadin)For Anticoagulation
Brief Title: Prospective Genotyping For Total Hip or Knee Replacement Patients Receiving Warfarin (Coumadin)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gwen McMillin (Other)
Responsible Party: Sponsor-Investigator, Gwen McMillin, Medical Director Toxicology and Trace Minterals, Department of Pathology, ARUP Laboratories, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00019469
Record Dates: First submitted 2008-02-06; First posted 2008-03-13 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-04

CONDITIONS: Venous Thromboembolism; Bleeding
Keywords: Genotyping; Warfarin dosing; arthroplasty
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacogenetic-based warfarin dosing (Experimental): Pharmacogenetic-based warfarin dosing: Warfarin dosing based on formula that incorporates genetic testing results.
  NOTE: Standard of care for elective knee and hip replacement at our institution is to receive post-operative warfarin thromboprophylaxis. Administration of warfarin was not specific to this study, nor was the duration of prophylaxis, however, warfarin dosing was influenced by the study arm, as noted above.
  Interventions: Genetic: Pharmacogenetic-based warfarin dosing
- Standard of care (control) (Active Comparator): Control or "usual care" warfarin dosing
  NOTE: Standard of care ("usual care") for elective knee and hip replacement at our institution is to receive post-operative warfarin thromboprophylaxis. Administration of warfarin was not specific to this study, nor was the duration of prophylaxis, however, warfarin dosing was influenced by the study arm, as noted above.
  Interventions: Other: Usual care warfarin dosing

INTERVENTIONS:
Genetic: Pharmacogenetic-based warfarin dosing — Prior to elective joint replacement surgery a blood sample is collected for genetic information(genotyping)which was used for calculating warfarin doses for patients randomized to the cytochrome arm. Outcomes in terms of efficacy, safety, and management of warfarin were compared between this group and the group in which warfarin doses are determined per usual care.
  NOTE: Standard of care for elective knee and hip replacement at our institution is to receive post-operative warfarin thromboprophylaxis. Administration of warfarin was not specific to this study, nor was the duration of prophylaxis, however, warfarin dosing was influenced by the study arm as noted above.
  Arms: Pharmacogenetic-based warfarin dosing
Other: Usual care warfarin dosing — For patients in arm 2, the control group, warfarin dosing is per usual care. Outcomes in terms of safety, efficacy, and warfarin management was compared to that of patients in the other arm, who receive warfarin dosing based on genotyping.
  NOTE: Standard of care for elective knee and hip replacement at our institution is to receive post-operative warfarin thromboprophylaxis. Administration of warfarin was not specific to this study, nor was the duration of prophylaxis, however, warfarin dosing was influenced by the study arm as noted above.
  Arms: Standard of care (control)

SUMMARY:
Several human genes affect how medications are metabolized by the body. It is believed that knowledge of variations of these genes can help health care providers better manage an anticoagulation medicine called warfarin (Coumadin®)and as a result decrease patient problems with bleeding or the development of blood clots. This study was designed to evaluate if genetic testing can improve warfarin initiation better than usual care.

DETAILED DESCRIPTION:
This study was completed in 2008 and was published. Consult the citation link for more details.

ELIGIBILITY:
Inclusion Criteria:

* Participants were otherwise healthy adults (≥ 18 years of age) who were planning total hip or knee replacement or revision surgery at the University of Utah Hospital, and scheduled a pre-operative office visit at the University of Utah Orthopaedic Center.

Exclusion Criteria:

* Blood transfusion in previous two weeks
* Participant is already taking warfarin
* Pre-operative INR > 4.0
* Pre-operative bilirubin > 2.4 mg/dL
* Current active cancer diagnosis with ongoing treatment
* Concomitant medications known to exert a major interaction with warfarin such as septra, metronidazole, tramadol, amiodarone, ciprofloxacin, or cimetidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwen McMillin, PhD, Principal Investigator — ARUP Laboratories
Locations (1):
- University of Utah Health Care, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McMillin GA, Melis R, Wilson A, Strong MB, Wanner NA, Vinik RG, Peters CL, Pendleton RC. Gene-based warfarin dosing compared with standard of care practices in an orthopedic surgery population: a prospective, parallel cohort study. Ther Drug Monit. 2010 Jun;32(3):338-45. doi: 10.1097/FTD.0b013e3181d925bb. PMID 20386359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients planning total hip or knee replacement surgery at the University of Utah Hospital, will be approached about participation in the study by Dr Chris Peters, MD or assigned orthopedic staff at the pre-operative office visit at the University of Utah Orthopaedic Center. Patients were enrolled from 9/27/06 - 10/2/08
Pre-assignment Details: Exclusion Criteria:
  1. Blood transfusion in previous two weeks
  2. Participant is already taking warfarin
  3. Pre-operative INR > 4.0
  4. Pre-operative bilirubin > 2.4 mg/dL
  5. Current active cancer diagnosis with ongoing treatment
  6. Concomitant medications known to exert a major interaction with warfarin
Groups:
- 2 Genotype Arm: The initial dose of warfarin will be corrected by the AC services team to account for variant genotypes, according to the following:
  Sqrt (Dose) = 0.628 - 0.0135(Age) - 0.240(CYP2C9*2) - 0.370 (CYP2C9*3) - 0.241(VKORC1) + 0.0162(Height) Age: input age in years CYP2C9: input 0, 1, or 2 based on the number of variant alleles VKORC1: input 1 for GG, 2 for GA, and 3 for AA Height: input height in centimeters Patients in this study group will be managed by designated AC services physicians, different from those in managing patients in the Control Arm of this study. Dosing adjustments will be made based on post-surgical INR values obtained initially on POD#2 daily during hospital stay, and 2 times weekly, or as needed, thereafter.
- 1 Control Arm: This is a two-armed parallel study with randomized assignment designed to test the hypothesis that selection of the initial warfarin dose based on CYP2C9 and VKORC1 genotypes will improve warfarin pharmacotherapy outcomes. Initial dose of warfarin will be given as per standard protocol for the Control Arm. Briefly, 3 or 5 mg warfarin will be administered on the day of surgery (post-operative day zero, POD#0) and the subsequent day. Patients in this study group will be managed by designated AC services physicians. Dosing adjustments will be made based on post-surgical INR values obtained initially on POD#2, daily during hospital stay, and 2 times weekly, or as needed, thereafter.
Period: Overall Study
Arm/Group | 2 Genotype Arm | 1 Control Arm
Started | 131 | 132
Completed | 114 | 115
Not Completed | 17 | 17
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 3 | 9
Not completed — Withdrawal by Subject | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Genotype-Based Dosing Arm: Initial warfarin dose calculated according to published Sconce algorithm
- Control Arm: Standard of care dosing
- Total: Total of all reporting groups
Arm/Group | Genotype-Based Dosing Arm | Control Arm | Total
Number analyzed (Participants) | 114 | 115 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 80 | 158
  >=65 years | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.18 (12.14) | 59.25 (12.83) | 58.75 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 72 | 140
  Male | 46 | 43 | 89
Region of Enrollment [Number; unit: participants]
  United States | 114 | 115 | 229

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events Associated With Warfarin Anticoagulation Following Total Hip and Total Knee Replacement
Description: Adverse events were defined as
  1. Major bleeding: fatal bleeding, bleeding into a critical organ, bleeding that requires hospital admission
  2. Minor bleeding: clinically overt bleeding not meeting criteria for major bleeding
  3. Symptomatic deep vein thrombosis (DVT)
  4. Pulmonary embolism (PE)
Time Frame: 90 days post surgery
Measure: Number; unit: participants
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
participants | 2 | 4

2. Secondary Outcome: Percentage of Determinations in Therapuetic Range (INR 1.8-2.9)
Description: Patient response to warfarin was evaluated based on the international normalized ratio (INR), calculated from a prothrombin time blood test. When the INR value was between 1.8 and 2.9, the patient was considered to be "therapeutic." The proportion of INR determinations that fell within the therapeutic range (INR between 1.8-2.9) was calculated, per arm, based on total number of INR determinations that were made during treatment with warfarin.
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hip arthroplasty)
Population: Determinations were assessed cumulatively throughout the study period, per patient, per arm. The total number of determinations was 804 for the genotype arm and 780 for the control arm
Measure: Number; unit: percentage of therapeutic INR values
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
percentage of therapeutic INR values | 43.3 | 44.9

3. Secondary Outcome: Percentage of Determinations Subtherapeutic (INR<1.8)
Description: Patient response to warfarin was evaluated based on the international normalized ratio (INR), calculated from a prothrombin time blood test. When the INR value was less than 1.8, the patient was considered to be "subtherapeutic." The proportion of INR determination that were subtherapeutic was caluculated, per arm, based on the total number of INR determinations that were made during treatment with warfarin.
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hop arthroplasty)
Population: as for outcome 2
Measure: Number; unit: percentage of deteminations
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
percentage of deteminations | 48.0 | 47.1

4. Secondary Outcome: Percentage of Determinations Supratherapeutic (INR>2.9)
Description: Patient response to warfarin was evaluated based on the international normalized ratio (INR), calculated from a prothrombin time blood test. When the INR value was greater than 2.9, the patient was considered to be "supratherapeutic." The proportion of INR determinations that were supratherapeutic was calculated, per arm, based on total number of INR determinations that were made during treatment with warfarin.
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hip arthroplasty)
Population: as for outcome 2
Measure: Number; unit: percentage of determinations
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
percentage of determinations | 8.7 | 8.0

5. Post Hoc Outcome: Mean Number of Doses Before First Dose Adjustment
Description: The number of consistent doses administered before the first dose adjustment was required was recorded, per patient. The average number of doses administered before the first dose adjustment is shown.
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hip arthroplasty)
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
doses | 3.1 (1.1) | 3.6 (1.3)

6. Post Hoc Outcome: Mean Number of Dose Adjustments
Description: The average number of dose adjustments made per patient, per arm, during the study period was calculated
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hip arthroplasty)
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
doses | 8.4 (2.18) | 7.0 (2.48)

7. Post Hoc Outcome: Percent of Patients With Dose Adjustments
Description: The percent of patients that required a dose adjustment during the study period was calculated.
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hip arthroplasty)
Measure: Number; unit: percentage of patients
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
percentage of patients | 83.5 | 78.0

8. Post Hoc Outcome: Mean Number of Doses Required for the First Therapeutic INR
Description: The number of doses required to achieve a therapeutic INR (1.8-2.9) was determined per patient, per arm. The average was then calculated and is shown here.
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hip arthroplasty)
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
doses | 3.9 (1.3) | 3.4 (1.1)

9. Post Hoc Outcome: Mean Number of Doses Before the First Supratherapeutic INR
Description: The number of warfarin doses administered before a patient INR exceeded the therapeutic range (>2.9) was recorded. The average was then calculated and is shown here.
Time Frame: 2 weeks (knee arthroplasty) or 4 weeks (hip arthroplasty)
Measure: Mean (Standard Deviation); unit: doses administered
Arm/Group | 2 Genotype Arm | 1 Control Arm
Number analyzed (Participants) | 114 | 115
doses administered | 5.4 (2.1) | 4.8 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded and investigated as they occurred, throughout the study period.
Arm/Group | 2 Genotype Arm | 1 Control Arm
Serious Adverse Events (participants affected / at risk) | 2/114 | 4/115
Other Adverse Events (participants affected / at risk) | 1/114 | 6/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Genotype Arm (N=114) | 1 Control Arm (N=115)
Venous thromboembolic event or bleed (Vascular disorders) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Genotype Arm (N=114) | 1 Control Arm (N=115)
Minor bleed (Vascular disorders) | 1 (1) | 6 (6) — Minor bleeds did not require hospitalization

LIMITATIONS AND CAVEATS:
Limited by the fact that INR was used to adjust dose at the third dose, which may not have allowed enough time for steady-state concentrations of warfarin to be achieved, nor for the genotype-based dosing to be adequately studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No